CLINICAL TRIAL: NCT04596644
Title: Impact of Repeatedly-Administered THC-cannabis on Experimental Pain and Abuse Liability in Humans
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: In response to quality assurance and compliance concerns, OHRP issued an FWA restriction on NYSPI research that included a pause of human research as of June 23, 2023.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Caroline A. Arout, Ph.D., Assistant Professor of Clinical Neurobiology (in Psychiatry), New York State Psychiatric Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8058; R21DA050752 (NIH)
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cannabis; Pain; Tolerance; Hyperalgesia
MeSH Terms: conditions — Marijuana Abuse; Pain; Hyperalgesia

STUDY DESIGN:
Intervention Model Description: This study comprises a 16-day inpatient stay. On the first full inpatient day (Day 1), participants will smoke one specified strength (Dose A) of cannabis. Days 2-8 will comprise Phase 1, in which a second strength (Dose B) of cannabis will be administered 3x/day. The next 7 days (Day 9-15) will be Phase 2, in which cannabis Dose A will be administered once again, at the same 3 daily time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose A: Standardization Phase (Experimental): On the first full inpatient day (Day 1), participants smoke one specified strength (Dose A; 75% of two 6.58% cannabis cigarettes) of cannabis at three timepoints.
  Interventions: Drug: Active Cannabis
- Dose B: Placebo Phase (Placebo Comparator): On Days 2-8, participants smoke a second strength (Dose B; 75% of two < 0.01%THC:CBD cannabis cigarettes) of cannabis will be administered 3x/day.
  Interventions: Drug: Placebo Cannabis
- Dose A: Active Phase (Experimental): On Days 9-15, cannabis Dose A will be administered again (75% of two 6.58% cannabis cigarettes) at three timepoints each day.
  Interventions: Drug: Active Cannabis

INTERVENTIONS:
Drug: Active Cannabis — 6.58% THC + <0.01% CBD cannabis (in one cigarette)
  Arms: Dose A: Active Phase; Dose A: Standardization Phase
Drug: Placebo Cannabis — <0.01% THC:CBD cannabis.
  Arms: Dose B: Placebo Phase

SUMMARY:
Chronic pain is a significant public health concern in the U.S., for which prescription opioids have historically been the standard treatment. This has resulted in striking rates of opioid use disorders and fatal overdoses. Identifying non-opioid medications for the management of chronic pain with minimal abuse liability is a public health necessity, and cannabinoids are a promising drug class for this purpose. More than 80% of medicinal cannabis users report pain as their primary medical indication, and they report experiencing minimal psychoactive effects. However, there are few well-controlled human laboratory studies assessing cannabis' efficacy for pain in the context of abuse, and even less is known regarding the effects of daily repeated use of cannabis on pain and its relationship to abuse liability. Carefully controlled research is needed.

The proposed randomized, within-subjects, placebo-controlled 16-day crossover inpatient human laboratory study (N = 20 healthy cannabis users; 10 men, 10 women) will address three important gaps in our understanding of the potential therapeutic utility of cannabis for pain: 1) Does tolerance develop to repeated, daily smoked cannabis administration on measures of experimental pain and abuse liability; 2) If so, is tolerance reversed during the 7 days of abstinence from active-THC cannabis; 3) Does abrupt abstinence from active cannabis increase experimental pain sensitivity, i.e. hyperalgesia, relative to baseline, and do these effects parallel measures of cannabis withdrawal such as disrupted mood and sleep?

Two distinct modalities of experimental pain will be assessed: The Cold Pressor Test (CPT) and Quantitative Sensory Testing Thermal Temporal Summation (QST-TTS). Throughout the study, experimental pain and abuse-related effects will be assessed, as will sleep and subjective mood assessments.

ELIGIBILITY:
Inclusion Criteria:

* Males/non-pregnant females, 21-60 years old
* Current cannabis user
* Able to perform all study procedures

Exclusion Criteria:

* Use of other illicit drugs
* If medical history, physical and psychiatric examination, or laboratory tests performed during the screening process reveal any significant illness that the study physician deems contraindicated for study participation
* Insensitivity to the cold-water stimulus of the Cold Pressor Test or the heat stimulus of Quantitative Sensory Testing

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cold Pressor Test (CPT) latency | Up to 15 days
  The CPT apparatus consists of two refrigerated circulators, filled with warm (36.5-37.5°C). participants will complete the CPT 30 minutes before the 1000h cannabis administration (baseline), and 0, 15, 30, 45, 60, and 90 minutes post-cannabis administration. and cold (3.5 - 4.5°C) water. Participants will insert their non-dominant hand into the warm water and remove it after 3 minutes; skin temperature of the thumb pad will be measured. Participants will then insert their hand in the cold water and will be instructed to report when they first experience pain (pain threshold) and remove their hand when the cold water can no longer be tolerated (pain tolerance). Maximum immersion time will be 3 minutes. Repeats on days 1, 2, 5, 8, 9, 12, and 15.

SECONDARY OUTCOMES:
Change in Quantitative Sensory Testing-Thermal Temporal Summation (QST-TTS) ratings | Up to 15 days
  The QST-TTS apparatus is a thermal testing analyzer with a 30 x 30 mm Peltier thermode, which will use repetitive nociceptive heat stimulation of a fixed frequency and intensity. At the beginning of the procedure, a research assistant (same gender as the participant) will read a script describing the procedure to the participant. Tonic noxious heat stimulation will be applied to the palm using a ramp-and-hold method, in which the baseline temperature will be set at 32.0°C, and will increase at a rate of 1°C/s up to 46.5°C, remaining constant for 120 sec. During the total duration of stimulation (135 seconds), participants will continuously rate the magnitude of perceived pain using a visual analog scale. participants will complete the CPT 30 minutes before the 1000h cannabis administration (baseline), and 0, 15, 30, 45, 60, and 90 minutes post-cannabis administration. Repeats on days 1, 2, 5, 8, 9, 12, and 15.
Change in Cannabis Rating Form (CRF) ratings | Up to 15 days
  Participants rate the strength, liking, desire to take again, good drug effect and bad. 7x on each of drug effect of cannabis on a 100mm visual analog scale. Repeats on days 1, 2, 5, 8, 9, 12, and 15.

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided